CLINICAL TRIAL: NCT05236257
Title: A Comparison of Clinical Outcomes in Infantile Fibrosarcoma (IFS) Patients Treated With Larotrectinib in the Phase I/II SCOUT Study Versus (an) External Historical Cohort(s)
Brief Title: A Study Called EPI VITRAKVI to Compare Treatment Results in Patients With Infantile Fibrosarcoma (IFS), a Type of Connective Soft Tissue Cancer, Who Received a Treatment Called Larotrectinib From a Study Called SCOUT With Patient Data From an External Database
Acronym: EPI VITRAKVI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21767
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced or Metastatic Infantile Fibrosarcoma Harboring an NTRK Gene Fusion; Infantile Fibrosarcoma
Keywords: Advanced solid tumors; Infantile fibrosarcoma (IFS); Neurotrophic tyrosine receptor kinase (NTRK); Fusion Positive; Tropomyosin Receptor Kinase (TRK) fusion; Larotrectinib; External control
MeSH Terms: interventions — larotrectinib; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Larotrectinib: Pediatric patients with IFS harboring an NTRK gene fusion who have been enrolled in the SCOUT study.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Standard care: Pediatric patients with IFS harboring an NTRK gene fusion in the eligible external cohort(s).
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Larotrectinib (Vitrakvi, BAY2757556) — Pediatric patients with IFS harboring an NTRK gene fusion.
  Groups: Larotrectinib
Drug: Standard of Care — Standard of care for the patients from the eligible external cohorts.
  Groups: Standard care

SUMMARY:
This is an observational study in which data from the past of children and young people with a specific cancer, called NTRK gene fusion positive infantile fibrosarcoma (IFS) is studied.

IFS is a rare type of childhood cancer that commonly affects legs and arms. IFS cancers typically have specific changes in their building plans (genes) called NTRK gene fusion. NTRK stands for the specific gene that has been altered, the neurotrophic tyrosine kinase (NTRK) gene.

This change to the building plan leads to the creation of an altered protein known as a TRK fusion protein, which can cause cancer cells to grow and to survive. The specific cancer is therefore also called TRK (tropomyosin receptor kinase) fusion-positive IFS.

The study drug, larotrectinib (also called BAY2757556) works by blocking the altered TRK fusion protein. Larotrectinib is already available in Europe and in many other countries and is approved for doctors to prescribe to patients with NTRK gene fusion cancer which has spread to nearby tissues and/or lymph nodes or to other parts of the body.

In France, HAS (the French authority in charge of evaluating health products and technologies) gave a positive opinion for the reimbursement of larotrectinib but only in the pediatric patients with IFS or another STS harboring a NTRK gene fusion, which is locally advanced or metastatic, and refractory or in relapse mainly due to the lack of comparative evidence.

The main purpose of this study is to collect more data to learn how well larotrectinib works compared with current standard of care chemotherapy in people up to 21 years of age with NTRK gene fusion positive IFS that has spread to nearby tissues and/or lymph nodes (locally advanced) or other parts of the body (metastatic).

To see how well larotrectinib works, researchers will make a comparison between

* how long larotrectinib works well and
* how long the standard of care works well.

Working well means that the treatments can prevent the following from happening:

* need for a new treatment for the cancer
* need for radiation therapy for the cancer
* need for surgery to treat the cancer, but which causes major damage to body parts
* death.

In addition to the above, data about medical problems related to the treatments in both groups and that may have required to stop the treatment will be compared.

The data for the comparison will come from

* an ongoing international study called SCOUT which was started in December 2015 (larotrectinib group)
* international databases (standard of care chemotherapy group). Data will be from the year 2000 up to the present.

There will be no required visits with a study doctor or required tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 21 years old.
* Locally advanced or metastatic Infantile Fibrosarcoma (IFS).
* Identification of an NTRK gene fusion by a molecular biology assay.
* Patients with available information on clinical, radiological characteristics of their tumor, therapies administered and outcomes.
* Patients receiving larotrectinib in the SCOUT trial.
* Patients receiving at least chemotherapy drugs in the historical control cohort(s).
* No opposition from the patients and/or representatives for data use.

Exclusion Criteria:

* Patients treated with TRK inhibitors in the historical control cohort(s).
* Patients with documented absence of NTRK gene fusion.
* Patients participating in an investigational program with interventions outside of routine clinical practice.

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population comprises of all pediatric patients in the SCOUT study and the eligible historical cohort(s) with a diagnosis of locally advanced or metastatic IFS harboring an NTRK gene fusion.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Carton M, Del Castillo JP, Colin JB, Kurtinecz M, Feuilly M, Pierron G, Arvis P, Khadir SK, Sparber-Sauer M, Orbach D. Larotrectinib versus historical standard of care in patients with infantile fibrosarcoma: protocol of EPI-VITRAKVI. Future Oncol. 2023 Aug;19(24):1645-1653. doi: 10.2217/fon-2023-0114. Epub 2023 May 3. PMID 37133249
- See also: VITRAKVI Patient Information — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=21767&attachmentIdentifier=ecffefac-d54c-4afb-9c04-46093c1d3330&fileName=21767_Patient_Information_Sheet_2.0.pdf&versionIdentifier=
- See also: Click here to find information for studies related to Bayer products. To find this study enter the NCT number or Bayer Study ID in the search field. — http://clinicaltrials.bayer.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted between 10-Mar-2022 (start retrospective observational study) and 13-Sep-2022 (table listing filles final) using secondary data.
  Three data sources were used in the study including SCOUT study (18 countries worldwide including France) and external historical control cohorts from the Institut Curie database and the Cooperative Weichteilsarkom Studiengruppe (CWS) database.
Pre-assignment Details: In total, 93 patients were included in this study (IFS population). The larotrectinib arm of the study included 51 patients from the SCOUT study. The single comparator arm of patients that received conventional chemotherapy included in total 42 external control patients, pooled from the Institut Curie database (N=18) and the CWS database (N=24).
Groups:
- Larotrectinib: Pediatric patients (up to 21 years old) with Infantile fibrosarcoma (IFS) harboring an NTRK gene fusion who have been enrolled in the SCOUT study (Bayer Study ID: 20290; NCT02637687) and treated with larotrectinib.
- External Controls: External historical control patients treated with at least one chemotherapy-based regimen, pooled from the Institut Curie (CURIE) database (N=18) and the Cooperative Weichteilsarkom Studiengruppe (CWS) database (N=24).
Period: Overall Study
Arm/Group | Larotrectinib | External Controls
Started | 51 | 42
Completed | 0 | 0
Not Completed | 51 | 42
Not completed — Ongoing with study treatment | 29 | 1
Not completed — Discontinued study treatment | 22 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Larotrectinib | External Controls | Total
Number analyzed (Participants) | 51 | 42 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.01 (3.49) | 0.73 (1.81) | 1.43 (2.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 30 | 27 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 51 | 42 | 93

OUTCOME MEASURES:

1. Primary Outcome: Time to Medical Treatment Failure
Description: Time to medical treatment failure was defined as the time (months) from the start of treatment to the date of the earliest event from: subsequent systemic treatment, radiation therapy, mutilating surgery or death due to any cause.
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
months
  Unweighted sample | NA [NA to NA] — median time to medical treatment failure was not estimable due to censored data | NA [57.1 to NA] — median time to medical treatment failure was not estimable due to censored data
  Weighted sample | NA [NA to NA] — median time to medical treatment failure was not estimable due to censored data | 24.0 [3.0 to NA] — upper limit of median time to medical treatment failure was not estimable due to censored data
Statistical Analysis 1: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.0058, Cox Proportional Hazards model; Unweighted; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.07 to 0.63]
Statistical Analysis 2: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.0023, Log Rank; Unweighted

2. Secondary Outcome: Time to Subsequent Systemic Treatment
Description: Time to subsequent systemic treatment was defined as the time from start date of Larotrectinib (for SCOUT) or start date of chemotherapy (for historical control cohorts) till the start date of a post-treatment systemic anti-cancer therapy, if any
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
months
  Unweighted Sample | NA [NA to NA] — median time to subsequent systemic treatment was not estimable due to censored data | NA [13.0 to NA] — median time to subsequent systemic treatment was not estimable due to censored data
  weighted Sample | NA [NA to NA] — median time to subsequent systemic treatment was not estimable due to censored data | 24.0 [24.0 to NA] — Upper limit of median time to subsequent systemic treatment was not estimable due to censored data
Statistical Analysis 1: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.0703, Cox Proportional Hazards model; Unweighted; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.05 to 1.13]
Statistical Analysis 2: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.0486, Log Rank; Unweighted

3. Secondary Outcome: Time to Mutilating Surgery Including Limb Amputation
Description: Time to mutilating surgery including limb amputation was defined as the time from start date of Larotrectinib (for SCOUT) or start date of chemotherapy (for historical control cohorts) till the start date of a mutilating surgery (including limb amputation)
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
months
  Unweighted Sample | NA [NA to NA] — median time to mutilating surgery including limb amputation was not estimable due to censored data | NA [NA to NA] — median time to mutilating surgery including limb amputation was not estimable due to censored data
  Weighted Sample | NA [NA to NA] — median time to mutilating surgery including limb amputation was not estimable due to censored data | NA [NA to NA] — median time to mutilating surgery including limb amputation was not estimable due to censored data
Statistical Analysis 1: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.696, Cox Proportional Hazards model; Unweighted; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.05 to 1.12]
Statistical Analysis 2: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.0476, Log Rank; Unweighted

4. Secondary Outcome: Time to First Radiation Therapy
Description: Time to radiation therapy was defined as the time from start date of Larotrectinib (for SCOUT) or start date of chemotherapy(for historical control cohorts) till the start date of a radiation therapy, if any
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
months
  Unweighted Sample | NA [NA to NA] — median time to first radiation therapy was not estimable due to censored data | NA [NA to NA] — median time to first radiation therapy was not estimable due to censored data
  Weighted Sample | NA [NA to NA] — median time to first radiation therapy was not estimable due to censored data | NA [NA to NA] — median time to first radiation therapy was not estimable due to censored data

5. Secondary Outcome: Time to Complete Surgical Resection
Description: Time to complete surgical resection (excluding amputation) was defined as the time from start date of Larotrectinib (for SCOUT) or start date of chemotherapy (for historical control cohorts) till the start date of a complete surgical resection (excluding amputation), if any
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
months
  Unweighted Sample | NA [NA to NA] — median time to complete surgical resection was not estimable due to censored data | NA [NA to NA] — median time to complete surgical resection was not estimable due to censored data
  Weighted Sample | NA [NA to NA] — median time to complete surgical resection was not estimable due to censored data | 6.1 [5.1 to NA] — upper limit of median time to complete surgical resection was not estimable due to censored data
Statistical Analysis 1: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.5713, Cox Proportional Hazards model; Unweighted; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.36 to 1.77]
Statistical Analysis 2: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.5695, Log Rank; Unweighted

6. Secondary Outcome: Overall Survival
Description: Number of participants with death due to any cause, alive, or lost to follow-up.
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Count of Participants; unit: Participants
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
Participants
  Dead | 1 | 3
  Alive | 50 | 39
Statistical Analysis 1: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.3200, Cox Proportional Hazards model; Unweighted; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.03 to 3.06]
Statistical Analysis 2: Comparison: Larotrectinib vs External Controls; Test type: Other; p = 0.2940, Log Rank; Unweighted

7. Secondary Outcome: Number of Participants With Treatment Discontinuation Due to Treatment Emergent Adverse Events
Description: Larotrectinib treatment for the SCOUT study and chemotherapy (first line) for the external historical control cohort(s).
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Measure: Count of Participants; unit: Participants
Arm/Group | Larotrectinib | External Controls
Number analyzed (Participants) | 51 | 42
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: up to 5.5 years for participants in SCOUT study and 22.5 years for participants in external historical control
Description: As it was stated in the protocol of the study, this retrospective observational study used secondary data collection from a previous clinical trial (SCOUT study) and from eligible databases used to select external historical control cohorts. Therefore, no new AEs or adverse drug reactions occurred besides the ones already described during the conduct of the initial clinical trial.
Arm/Group | Larotrectinib | External Controls
All-Cause Mortality (participants affected / at risk) | 1/51 | 3/42
Serious Adverse Events (participants affected / at risk) | 1/51 | 3/42
Other Adverse Events (participants affected / at risk) | 0/51 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Larotrectinib (N=51) | External Controls (N=42)
Death (General disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure agreement is that the publication is restricted for external partners.

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05236257/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT05236257/SAP_001.pdf